CLINICAL TRIAL: NCT03875651
Title: A U.S. Post-Approval Study of the SYNERGY 4.50/5.00 mm Everolimus-Eluting Platinum Chromium Coronary Stent System (Evolve 4.5/5.0)
Brief Title: A Clinical Trial to Confirm Safety & Effectiveness of the SYNERGY 4.50 mm and 5.00 mm Stent for Treatment of Atherosclerotic Lesion(s)
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2357
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Atherosclerosis; Heart Diseases, Coronary; Coronary Artery Disease; Cardiovascular Diseases
Keywords: Drug-Eluting Stents
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: SYNERGY 4.50 mm and 5.0 mm Coronary Stent System — The SYNERGY Everolimus-Eluting Platinum Chromium Coronary Stent System (SYNERGY Stent System), manufactured by BSC, is a device/drug combination product comprised of two regulated components: a device (Coronary Stent System) and a drug product (a formulation of everolimus contained in a bioabsorbable polymer coating).

SUMMARY:
EVOLVE 4.5/5.0 is a prospective, single-arm, multi-center observational (standard of care) trial intended to confirm the safety and effectiveness of the SYNERGY 4.50 mm and 5.00 mm Coronary Stent System for the treatment of patients with coronary artery disease in large vessels (≤ 28 mm in length, by visual estimate, in native coronary arteries > 4.00 mm to ≤5.00 mm in diameter, by visual estimate). This Post Approval study is a cohort associated with the SYNERGY MEGATRON Post Approval Study, which is registered under ClinicalTrials.gov ID: NCT04807439.

ELIGIBILITY:
Inclusion Criteria:

* A patient is an acceptable candidate if they require treatment with a 4.50 or 5.00 mm SYNERGY stent for the treatment of their disease in accordance with the applicable guidelines on PCI, the SYNERGY DFU, and the Declaration of Helsinki.

Exclusion Criteria:

* Planned treatment with a non-SYNERGY stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients include those with atherosclerotic coronary lesions with vessel diameters that can appropriately be treated with 4.50 mm and/or 5.00 mm stents according to the commercially approved SYNERGY DFU
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) rate | 12-months
  12-month Target Lesion Failure (TLF) rate, defined as any ischemia driven revascularization of the target lesion (TLR), myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel, or cardiac death.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Stoler, MD, Principal Investigator — Baylor Heart and Vascular Hospital
Locations (9):
- United States (9):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - North Kansas City Hospital, Kansas City, Missouri
  - Wake Medical Center, Raleigh, North Carolina
  - Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - Oregon Health Science University, Portland, Oregon
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Inova Fairfax Hospital, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy: (http://www.bostonscientific.com/en-US/data-sharing-requests.html).